CLINICAL TRIAL: NCT06856161
Title: A Novel Blood Test as a Differential Diagnosis and Drug Efficacy Biomarker in Mental Health
Brief Title: A Novel Blood Test as a Biomarker in Mental Health
Acronym: LEADING-MH
Status: Not yet recruiting | Type: Observational
Sponsor: Steve Reynolds (Other)
Collaborators: Royal Columbian Hospital Foundation (Other)
Responsible Party: Sponsor-Investigator, Steve Reynolds, MD, FRCPC, Fraser Health
Organization: Fraser Health (Other)
Other Study IDs: FHREB 2024-143
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Depression - Major Depressive Disorder; Schizophenia Disorder; Psychosis; Mania (Neurotic); Alcohol Consumption; Anxiety Disorder (Panic Disorder or GAD); Substance Use Disorders; Alcohol Use Disorder
Keywords: mental health; biomarker; depression; schizophrenia; psychosis; SERT
MeSH Terms: conditions — Psychotic Disorders; Mania; Alcohol Drinking; Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder; Substance-Related Disorders; Alcoholism; Psychological Well-Being; Depression; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DEP: Participants with suspected, new-onset, or established depression presenting to the psychiatric outpatient clinic at Royal Columbian Hospital.
- PSY: Participants experiencing a first episode of psychosis or established schizophrenia presenting to an outpatient psychosis clinic at Royal Columbian Hospital.

SUMMARY:
This longitudinal, observational study aims to assess whether the characteristics of a novel blood peripheral biomarker can serve as indicators for depression and schizophrenia in patients at the Royal Columbian Hospital Psychiatric Clinics. The study will evaluate whether changes in these biomarker characteristics can help distinguish between depressed patients who do or do not respond to treatment and between individuals experiencing a single psychotic episode and those at risk of progressing to schizophrenia. To achieve this, blood samples and standardized mental health assessments will be collected across three study visits from up to 500 participants, grouped into two study arms based on their diagnosis: Depression (DEP) or Psychosis/Schizophrenia (PSY).

ELIGIBILITY:
Inclusion Criteria:

I. Age 19+. II. Informed consent by participant

III. Any of the following situations:

1. Suspected, new onset or established depression.
2. First episode of psychosis or suspected/established schizophrenia. IV. In the opinion of the Investigator, the participant will likely be able to complete the standardized mental health questionnaires administered in each study visit.

Exclusion Criteria:

I. Inability to provide informed consent. II. Currently enrolled in any other research study involving drugs or devices that may confound mental health treatment outcomes.

III. Currently declared on extended leave Under British Columbia's Mental Health Act.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 500 adults (19 years and older) with suspected or diagnosed Major Depressive Disorder (MDD) or psychotic disorders, including schizophrenia, who are receiving care at psychiatric clinics at Royal Columbian Hospital (RCH) in New Westminster, Canada. The study population will be diverse in age, gender, ethnicity, and socioeconomic background, reflecting the demographics of RCH patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Relationship between Depression and Biomarker Characteristics | 6 months from enrollment, across three study visits.
  In the DEP arm, the study will evaluate the relationship between depression diagnosis, antidepressant responsiveness (assessed through changes in a standardized mental health questionnaire over time), and the characteristics of a novel blood peripheral biomarker.
Relationship between Psychotic Disorders and Biomarker Characteristics | 6 months from enrollment, across 3 study visits.
  In the PSY arm, the study will evaluate the relationship between schizophrenia (defined as chronic, recurrent psychosis) and other psychotic disorders and the characteristics of a novel blood peripheral biomarker. A standardized clinical assessment tool will be used to support the diagnosis of schizophrenia.

SECONDARY OUTCOMES:
Association between Clinical-Demographic Factors and Biomarker Characteristics. | 6 months from enrollment, across 3 study visits.
  In the DEP arm, the study will evaluate the relationship between a novel blood peripheral biomarker and various clinical and demographic factors. These factors include time, age, sex assigned at birth, and symptom severity related to suicidality, anxiety, substance use, and inflammation. Standardized mental health and clinical assessment tools will be used to quantify these variables.
Relationship between PSY arm Clinical-Demographic Factors and Biomarker Characteristics. | 6 months from enrollment, across 3 study visits.
  In the PSY arm, the study will evaluate the relationship between the characteristics of a novel blood peripheral biomarker and various clinical and demographic factors. These factors include time, age, sex assigned at birth, and symptom severity related to psychosis, suicidality, anxiety, substance use, and inflammation. Standardized mental health and clinical assessment tools will be used to quantify these variables.
Association between Psychotic Disorders Pharmacological Treatment and Biomarker Characteristics | 6 months from enrollment, across 3 study visits.
  In the PSY arm, the study will evaluate the relationship between changes over time in the characteristics of a novel blood peripheral biomarker and exposure to antipsychotics and other non-SSRI medications.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, MD, FRCPC, Principal Investigator — Royal Columbian Hospital Foundation
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romay-Tallon R, Kulhawy E, Brymer KJ, Allen J, Rivera-Baltanas T, Olivares JM, Kalynchuk LE, Caruncho HJ. Changes in Membrane Protein Clustering in Peripheral Lymphocytes in an Animal Model of Depression Parallel Those Observed in Naive Depression Patients: Implications for the Development of Novel Biomarkers of Depression. Front Pharmacol. 2018 Oct 15;9:1149. doi: 10.3389/fphar.2018.01149. eCollection 2018. PMID 30374301
- [Background] Rodrigues-Amorim D, Rivera-Baltanas T, Lopez M, Spuch C, Olivares JM, Agis-Balboa RC. Schizophrenia: A review of potential biomarkers. J Psychiatr Res. 2017 Oct;93:37-49. doi: 10.1016/j.jpsychires.2017.05.009. Epub 2017 May 26. PMID 28578207
- [Background] Rivera-Baltanas T, Olivares JM, Martinez-Villamarin JR, Fenton EY, Kalynchuk LE, Caruncho HJ. Serotonin 2A receptor clustering in peripheral lymphocytes is altered in major depression and may be a biomarker of therapeutic efficacy. J Affect Disord. 2014 Jul;163:47-55. doi: 10.1016/j.jad.2014.03.011. Epub 2014 Apr 3. PMID 24836087
- [Background] Rivera-Baltanas T, Olivares JM, Calado-Otero M, Kalynchuk LE, Martinez-Villamarin JR, Caruncho HJ. Serotonin transporter clustering in blood lymphocytes as a putative biomarker of therapeutic efficacy in major depressive disorder. J Affect Disord. 2012 Mar;137(1-3):46-55. doi: 10.1016/j.jad.2011.12.041. Epub 2012 Jan 16. PMID 22257570
- [Background] Rivera-Baltanas T, Agis-Balboa RC, Romay-Tallon R, Kalynchuk LE, Olivares JM, Caruncho HJ. Serotonin transporter clustering in blood lymphocytes predicts the outcome on anhedonia scores in naive depressive patients treated with antidepressant medication. Ann Gen Psychiatry. 2015 Dec 21;14:45. doi: 10.1186/s12991-015-0085-8. eCollection 2015. PMID 26697099
- [Background] Rangaswamy T, Mangala R, Mohan G, Joseph J, John S. Intervention for first episode psychosis in India - The SCARF experience. Asian J Psychiatr. 2012 Mar;5(1):58-62. doi: 10.1016/j.ajp.2012.01.011. Epub 2012 Mar 3. PMID 26878950
- [Background] Peterson BS. Editorial: Biomarkers in precision medicine for mental illnesses. J Child Psychol Psychiatry. 2020 Dec;61(12):1279-1281. doi: 10.1111/jcpp.13357. PMID 33252151
- [Background] Orsolini L, Pompili S, Tempia Valenta S, Salvi V, Volpe U. C-Reactive Protein as a Biomarker for Major Depressive Disorder? Int J Mol Sci. 2022 Jan 30;23(3):1616. doi: 10.3390/ijms23031616. PMID 35163538
- [Background] Ormel J, Hollon SD, Kessler RC, Cuijpers P, Monroe SM. More treatment but no less depression: The treatment-prevalence paradox. Clin Psychol Rev. 2022 Feb;91:102111. doi: 10.1016/j.cpr.2021.102111. Epub 2021 Dec 11. PMID 34959153
- [Background] Obermeier M, Schennach-Wolff R, Meyer S, Moller HJ, Riedel M, Krause D, Seemuller F. Is the PANSS used correctly? a systematic review. BMC Psychiatry. 2011 Jul 18;11:113. doi: 10.1186/1471-244X-11-113. PMID 21767349
- [Background] National Collaborating Centre for Mental Health (UK). Psychosis and Schizophrenia in Adults: Treatment and Management: Updated Edition 2014. London: National Institute for Health and Care Excellence (UK); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK248060/ PMID 25340235
- [Background] Murphy SE, Capitao LP, Giles SLC, Cowen PJ, Stringaris A, Harmer CJ. The knowns and unknowns of SSRI treatment in young people with depression and anxiety: efficacy, predictors, and mechanisms of action. Lancet Psychiatry. 2021 Sep;8(9):824-835. doi: 10.1016/S2215-0366(21)00154-1. PMID 34419187
- [Background] Munkholm K, Winkelbeiner S, Homan P. Individual response to antidepressants for depression in adults-a meta-analysis and simulation study. PLoS One. 2020 Aug 27;15(8):e0237950. doi: 10.1371/journal.pone.0237950. eCollection 2020. PMID 32853222
- [Background] Moreno-Agostino D, Wu YT, Daskalopoulou C, Hasan MT, Huisman M, Prina M. Global trends in the prevalence and incidence of depression:a systematic review and meta-analysis. J Affect Disord. 2021 Feb 15;281:235-243. doi: 10.1016/j.jad.2020.12.035. Epub 2020 Dec 9. PMID 33338841
- [Background] Meyer TD, Crist N, La Rosa N, Ye B, Soares JC, Bauer IE. Are existing self-ratings of acute manic symptoms in adults reliable and valid?-A systematic review. Bipolar Disord. 2020 Sep;22(6):558-568. doi: 10.1111/bdi.12906. Epub 2020 Apr 13. PMID 32232950
- [Background] Howes OD, Egerton A, Allan V, McGuire P, Stokes P, Kapur S. Mechanisms underlying psychosis and antipsychotic treatment response in schizophrenia: insights from PET and SPECT imaging. Curr Pharm Des. 2009;15(22):2550-9. doi: 10.2174/138161209788957528. PMID 19689327
- [Background] McCutcheon RA, Pillinger T, Efthimiou O, Maslej M, Mulsant BH, Young AH, Cipriani A, Howes OD. Reappraising the variability of effects of antipsychotic medication in schizophrenia: a meta-analysis. World Psychiatry. 2022 Jun;21(2):287-294. doi: 10.1002/wps.20977. PMID 35524614
- [Background] McCutcheon RA, Pillinger T, Mizuno Y, Montgomery A, Pandian H, Vano L, Marques TR, Howes OD. The efficacy and heterogeneity of antipsychotic response in schizophrenia: A meta-analysis. Mol Psychiatry. 2021 Apr;26(4):1310-1320. doi: 10.1038/s41380-019-0502-5. Epub 2019 Aug 30. PMID 31471576
- [Background] Matson TE, Hallgren KA, Lapham GT, Oliver M, Wang X, Williams EC, Bradley KA. Psychometric Performance of a Substance Use Symptom Checklist to Help Clinicians Assess Substance Use Disorder in Primary Care. JAMA Netw Open. 2023 May 1;6(5):e2316283. doi: 10.1001/jamanetworkopen.2023.16283. PMID 37234003
- [Background] Maslej MM, Furukawa TA, Cipriani A, Andrews PW, Mulsant BH. Individual Differences in Response to Antidepressants: A Meta-analysis of Placebo-Controlled Randomized Clinical Trials. JAMA Psychiatry. 2020 Jun 1;77(6):607-617. doi: 10.1001/jamapsychiatry.2019.4815. PMID 32074273
- [Background] Maslej MM, Furukawa TA, Cipriani A, Andrews PW, Sanches M, Tomlinson A, Volkmann C, McCutcheon RA, Howes O, Guo X, Mulsant BH. Individual Differences in Response to Antidepressants: A Meta-analysis of Placebo-Controlled Randomized Clinical Trials. JAMA Psychiatry. 2021 May 1;78(5):490-497. doi: 10.1001/jamapsychiatry.2020.4564. PMID 33595620
- [Background] Kesby JP, Eyles DW, McGrath JJ, Scott JG. Dopamine, psychosis and schizophrenia: the widening gap between basic and clinical neuroscience. Transl Psychiatry. 2018 Jan 31;8(1):30. doi: 10.1038/s41398-017-0071-9. PMID 29382821
- [Background] Lappin JM, Heslin M, Lomas B, Jones PB, Doody GA, Reininghaus UA, Croudace T, Craig T, Fearon P, Murray RM, Dazzan P, Morgan C. Early sustained recovery following first episode psychosis: Evidence from the AESOP10 follow-up study. Schizophr Res. 2018 Sep;199:341-345. doi: 10.1016/j.schres.2018.03.014. Epub 2018 Mar 20. PMID 29571751
- [Background] Leichsenring F, Steinert C, Rabung S, Ioannidis JPA. The efficacy of psychotherapies and pharmacotherapies for mental disorders in adults: an umbrella review and meta-analytic evaluation of recent meta-analyses. World Psychiatry. 2022 Feb;21(1):133-145. doi: 10.1002/wps.20941. PMID 35015359
- [Background] Leighton SP, Nerurkar L, Krishnadas R, Johnman C, Graham GJ, Cavanagh J. Chemokines in depression in health and in inflammatory illness: a systematic review and meta-analysis. Mol Psychiatry. 2018 Jan;23(1):48-58. doi: 10.1038/mp.2017.205. Epub 2017 Nov 14. PMID 29133955
- [Background] Lenze EJ, Rodebaugh TL, Nicol GE. A Framework for Advancing Precision Medicine in Clinical Trials for Mental Disorders. JAMA Psychiatry. 2020 Jul 1;77(7):663-664. doi: 10.1001/jamapsychiatry.2020.0114. No abstract available. PMID 32211837
- [Background] Marasine NR, Sankhi S, Lamichhane R, Marasini NR, Dangi NB. Use of Antidepressants among Patients Diagnosed with Depression: A Scoping Review. Biomed Res Int. 2021 Mar 15;2021:6699028. doi: 10.1155/2021/6699028. eCollection 2021. PMID 33791379
- [Background] Kang HJ, Kim JW, Choi W, Lee JY, Kim SW, Shin IS, Kim JM. Use of Serum Biomarkers to Aid Antidepressant Selection in Depressive Patients. Clin Psychopharmacol Neurosci. 2024 Feb 29;22(1):182-187. doi: 10.9758/cpn.23.1071. Epub 2023 Jun 29. PMID 38247424
- [Background] Kadakia A, Catillon M, Fan Q, Williams GR, Marden JR, Anderson A, Kirson N, Dembek C. The Economic Burden of Schizophrenia in the United States. J Clin Psychiatry. 2022 Oct 10;83(6):22m14458. doi: 10.4088/JCP.22m14458. PMID 36244006
- [Background] Jackson-Koku G. Beck Depression Inventory. Occup Med (Lond). 2016 Mar;66(2):174-5. doi: 10.1093/occmed/kqv087. No abstract available. PMID 26892598
- [Background] Institute for Health Metrics and Evaluation. (2021). GBD Compare. Retrieved from IHME, University of Washington: https://vizhub.healthdata.org/gbd-compare/
- [Background] Higgins-Biddle JC, Babor TF. A review of the Alcohol Use Disorders Identification Test (AUDIT), AUDIT-C, and USAUDIT for screening in the United States: Past issues and future directions. Am J Drug Alcohol Abuse. 2018;44(6):578-586. doi: 10.1080/00952990.2018.1456545. Epub 2018 May 3. PMID 29723083
- [Background] Gutsmiedl K, Krause M, Bighelli I, Schneider-Thoma J, Leucht S. How well do elderly patients with major depressive disorder respond to antidepressants: a systematic review and single-group meta-analysis. BMC Psychiatry. 2020 Mar 4;20(1):102. doi: 10.1186/s12888-020-02514-2. PMID 32131786
- [Background] Gururajan A, Clarke G, Dinan TG, Cryan JF. Molecular biomarkers of depression. Neurosci Biobehav Rev. 2016 May;64:101-33. doi: 10.1016/j.neubiorev.2016.02.011. Epub 2016 Feb 21. PMID 26906761
- [Background] Guloksuz S, van Os J. The slow death of the concept of schizophrenia and the painful birth of the psychosis spectrum. Psychol Med. 2018 Jan;48(2):229-244. doi: 10.1017/S0033291717001775. Epub 2017 Jul 10. PMID 28689498
- [Background] Greenfield P, Joshi S, Christian S, Lekkos P, Gregorowicz A, Fisher HL, Johnson S. First episode psychosis in the over 35 s: is there a role for early intervention? Early Interv Psychiatry. 2018 Jun;12(3):348-354. doi: 10.1111/eip.12322. Epub 2016 Mar 28. PMID 27018640
- [Background] Greenberg P, Chitnis A, Louie D, Suthoff E, Chen SY, Maitland J, Gagnon-Sanschagrin P, Fournier AA, Kessler RC. The Economic Burden of Adults with Major Depressive Disorder in the United States (2019). Adv Ther. 2023 Oct;40(10):4460-4479. doi: 10.1007/s12325-023-02622-x. Epub 2023 Jul 31. PMID 37518849
- [Background] Felger JC, Haroon E, Patel TA, Goldsmith DR, Wommack EC, Woolwine BJ, Le NA, Feinberg R, Tansey MG, Miller AH. What does plasma CRP tell us about peripheral and central inflammation in depression? Mol Psychiatry. 2020 Jun;25(6):1301-1311. doi: 10.1038/s41380-018-0096-3. Epub 2018 Jun 12. PMID 29895893
- [Background] FDA-NIH Biomarker Working Group. BEST (Biomarkers, EndpointS, and other Tools) Resource [Internet]. Silver Spring (MD): Food and Drug Administration (US); 2016-. Available from http://www.ncbi.nlm.nih.gov/books/NBK326791/ PMID 27010052
- [Background] Eilert N, Enrique A, Wogan R, Mooney O, Timulak L, Richards D. The effectiveness of Internet-delivered treatment for generalized anxiety disorder: An updated systematic review and meta-analysis. Depress Anxiety. 2021 Feb;38(2):196-219. doi: 10.1002/da.23115. Epub 2020 Nov 22. PMID 33225589
- [Background] Crespo-Facorro B, Such P, Nylander AG, Madera J, Resemann HK, Worthington E, O'Connor M, Drane E, Steeves S, Newton R. The burden of disease in early schizophrenia - a systematic literature review. Curr Med Res Opin. 2021 Jan;37(1):109-121. doi: 10.1080/03007995.2020.1841618. Epub 2020 Nov 13. PMID 33095689
- [Background] Correll CU, Howes OD. Treatment-Resistant Schizophrenia: Definition, Predictors, and Therapy Options. J Clin Psychiatry. 2021 Sep 7;82(5):MY20096AH1C. doi: 10.4088/JCP.MY20096AH1C. PMID 34496461
- [Background] Charlson FJ, Ferrari AJ, Santomauro DF, Diminic S, Stockings E, Scott JG, McGrath JJ, Whiteford HA. Global Epidemiology and Burden of Schizophrenia: Findings From the Global Burden of Disease Study 2016. Schizophr Bull. 2018 Oct 17;44(6):1195-1203. doi: 10.1093/schbul/sby058. PMID 29762765
- [Background] Carvalho AF, Solmi M, Sanches M, Machado MO, Stubbs B, Ajnakina O, Sherman C, Sun YR, Liu CS, Brunoni AR, Pigato G, Fernandes BS, Bortolato B, Husain MI, Dragioti E, Firth J, Cosco TD, Maes M, Berk M, Lanctot KL, Vieta E, Pizzagalli DA, Smith L, Fusar-Poli P, Kurdyak PA, Fornaro M, Rehm J, Herrmann N. Evidence-based umbrella review of 162 peripheral biomarkers for major mental disorders. Transl Psychiatry. 2020 May 18;10(1):152. doi: 10.1038/s41398-020-0835-5. PMID 32424116
- [Background] Boyce P, Hopwood M, Morris G, Hamilton A, Bassett D, Baune BT, Mulder R, Porter R, Parker G, Singh AB, Outhred T, Das P, Malhi GS. Switching antidepressants in the treatment of major depression: When, how and what to switch to? J Affect Disord. 2020 Jan 15;261:160-163. doi: 10.1016/j.jad.2019.09.082. Epub 2019 Sep 30. PMID 31630037
- [Background] Biomarkers Definitions Working Group.. Biomarkers and surrogate endpoints: preferred definitions and conceptual framework. Clin Pharmacol Ther. 2001 Mar;69(3):89-95. doi: 10.1067/mcp.2001.113989. No abstract available. PMID 11240971
- [Background] American Psychiatric Association. (2024, April). What Is Depression? Retrieved from American Psychiatric Association: https://www.psychiatry.org/patients-families/depression/what-is-depression
- [Background] American Psychiatric Association. (2020, October). Schizophrenia. Retrieved from American Psychiatric Association: https://www.psychiatry.org/patients-families/schizophrenia
- [Background] Alvarez-Jimenez M, Gleeson JF, Henry LP, Harrigan SM, Harris MG, Amminger GP, Killackey E, Yung AR, Herrman H, Jackson HJ, McGorry PD. Prediction of a single psychotic episode: a 7.5-year, prospective study in first-episode psychosis. Schizophr Res. 2011 Feb;125(2-3):236-46. doi: 10.1016/j.schres.2010.10.020. Epub 2010 Nov 16. PMID 21081266
- [Background] Altman EG, Hedeker D, Peterson JL, Davis JM. The Altman Self-Rating Mania Scale. Biol Psychiatry. 1997 Nov 15;42(10):948-55. doi: 10.1016/S0006-3223(96)00548-3. PMID 9359982
- [Background] Abi-Dargham A, Moeller SJ, Ali F, DeLorenzo C, Domschke K, Horga G, Jutla A, Kotov R, Paulus MP, Rubio JM, Sanacora G, Veenstra-VanderWeele J, Krystal JH. Candidate biomarkers in psychiatric disorders: state of the field. World Psychiatry. 2023 Jun;22(2):236-262. doi: 10.1002/wps.21078. PMID 37159365